CLINICAL TRIAL: NCT05309902
Title: A Phase 1, Double-Blinded, Placebo- and Active-Controlled, Randomized Study to Investigate the Potential of Soticlestat to Prolong the QTc Interval in Healthy Adult Participants
Brief Title: A Study of Soticlestat in Healthy Adults To Evaluate the Effect on QTc Interval
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study not needed
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: TAK-935-1001
Record Dates: First submitted 2022-03-30; First posted 2022-04-04 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy
MeSH Terms: interventions — soticlestat; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Sequence 1: (Regimen A + Regimen B + Regimen C + Regimen D) (Experimental): Regimen A (soticlestat 300 milligram [mg] tablets + soticlestat placebo-matching tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition once on Day 1 of Treatment Period 1, followed by at least 7 days washout period, followed by Regimen B (soticlestat 900 mg tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition once on Day 1 of Treatment Period 2, followed by at least 7 days washout period, followed by Regimen C (soticlestat placebo-matching tablets + moxifloxacin 400 mg over-encapsulated tablet), orally, in fasting condition, once on Day 1 of Treatment Period 3, followed by at least 7 days washout period, followed by Regimen D (soticlestat placebo-matching tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition once on Day 1 of Treatment Period 4.
  Interventions: Drug: Soticlestat; Drug: Placebo; Drug: Moxifloxacin
- Sequence 2: (Regimen B + Regimen D + Regimen A + Regimen C) (Experimental): Regimen B (soticlestat 900 mg tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition once on Day 1 of Treatment Period 1, followed by at least 7 days washout period, followed by Regimen D (soticlestat placebo-matching tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition once on Day 1 of Treatment Period 2, followed by at least 7 days washout period, followed by Regimen A (soticlestat 300 mg tablets + soticlestat placebo-matching tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition, once on Day 1 of Treatment Period 3, followed by at least 7 days washout period, followed by Regimen C (soticlestat -matching tablets + moxifloxacin 400 mg over-encapsulated tablet), orally, in fasting condition once on Day 1 of Treatment Period 4.
  Interventions: Drug: Soticlestat; Drug: Placebo; Drug: Moxifloxacin
- Sequence 3: (Regimen C + Regimen A + Regimen D + Regimen B) (Experimental): Regimen C (soticlestat placebo-matching tablets + moxifloxacin 400 mg over-encapsulated tablet), orally, in fasting condition once on Day 1 of Treatment Period 1, followed by at least 7 days washout period, followed by Regimen A (soticlestat 300 mg tablets + soticlestat placebo-matching tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition once on Day 1 of Treatment Period 2, followed by at least 7 days washout period, followed by Regimen D (soticlestat placebo-matching tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition, once on Day 1 of Treatment Period 3, followed by at least 7 days washout period, followed by Regimen B (soticlestat 900 mg tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition once on Day 1 of Treatment Period 4.
  Interventions: Drug: Soticlestat; Drug: Placebo; Drug: Moxifloxacin
- Sequence 4: (Regimen D + Regimen C + Regimen B + Regimen A) (Experimental): Regimen D (soticlestat placebo-matching tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition once on Day 1 of Treatment Period 1, followed by at least 7 days washout period, followed by Regimen C (soticlestat placebo-matching tablets + moxifloxacin 400 mg over-encapsulated tablet), orally, in fasting condition once on Day 1 of Treatment Period 2, followed by at least 7 days washout period, followed by Regimen B (soticlestat 900 mg tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition, once on Day 1 of Treatment Period 3, followed by at least 7 days washout period, followed by Regimen A (soticlestat 300 mg tablets + soticlestat placebo-matching tablets + moxifloxacin placebo-matching capsule), orally, in fasting condition once on Day 1 of Treatment Period 4.
  Interventions: Drug: Soticlestat; Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Soticlestat — Soticlestat tablet.
  Other Names: TAK-935
Drug: Placebo — Soticlestat placebo-matching tablet.
Drug: Moxifloxacin — Moxifloxacin over-encapsulated tablet.
Drug: Placebo — Moxifloxacin placebo-matching capsule.

SUMMARY:
The main aim is to see if soticlestat has any effect in the heart rate.

Participants will receive 4 doses of soticlestat in tablets and will complete some assessment which include to record activity of the heart and collection of blood samples.

Then, the clinic will contact the participants 14 days after their final dose of soticlestat to check if they have any health problems.

DETAILED DESCRIPTION:
The drug being tested in this study is called soticlestat. Soticlestat is being tested in healthy participants for the purpose of this study. This study will assess the effect of single-dose of soticlestat on the heart rate (QTc prolongation). The study will enroll approximately 60 participants.

Participants will be randomly assigned (by chance, like flipping a coin) to 1 of the 4 treatments sequences.

* Sequence 1: (Regimen A+ Regimen B + Regimen C + Regimen D)
* Sequence 2: (Regimen B+ Regimen D + Regimen A + Regimen C)
* Sequence 3: (Regimen C+ Regimen A + Regimen D + Regimen B)
* Sequence 4: (Regimen D+ Regimen C + Regimen B + Regimen A)

All participants will receive all 4 treatment regimens. Treatment order will remain undisclosed to the participants and study doctor (unless there is an urgent medical need). This is a single-center trial. Participants will be followed up for up to 14 days after the last dose of study drug for a follow-up assessment. The overall time to participate in this study is approximately 63 days including screening period and follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Male participants agree to comply with any applicable contraceptive requirements of the protocol.
2. Body mass index (BMI) greater than or equal to (>=)18.0 and <=32.0 kilogram per square meter (kg/m^2) at screening.
3. Continuous non-smoker who has not used nicotine-containing products for at least 90 days prior to the first dosing, based on participant self-reporting.
4. No clinically significant history or presence of ECG findings as judged by the Investigator or designee, including each criterion as listed below:

   * Normal sinus rhythm (HR between 45 bpm and 100 bpm inclusive) at screening and check-in;
   * QTcF is <=450 ms (males) or <=470 ms (females) at screening and check-in;
   * QRS interval <=110 ms; if >110 ms, result will be confirmed by a manual over read at screening and check-in;
   * PR interval <=220 ms at screening and check-in.

Exclusion Criteria:

1. Mentally or legally incapacitated or has significant emotional problems at the time of the screening visit or expected during the conduct of the study.
2. History or presence of any of the following, deemed clinically significant by the Investigator or designee:

   * epilepsy, seizure, or convulsion, tremor or related symptoms;
   * risk factors for Torsade de Pointes (TdP) (example, heart failure, unexplained syncope, cardiomyopathy, or family history of Long QT Syndrome);
   * family history of sudden death;
   * sick sinus syndrome, second or third degree atrioventricular block, myocardial infarction, pulmonary congestion, symptomatic or significant cardiac arrhythmia, prolonged QTcF interval, or conduction abnormalities;
   * ischemic heart disease, poorly controlled hypertension, or other cardiovascular disorder;
   * T wave flattening or other abnormalities which in the opinion of the investigator or designee may interfere with the analysis of QT intervals;
   * clinically significant hyper- or hypokalemia.
3. Any positive responses on the Columbia-Suicide Severity Rating Scale (C-SSRS) that in the clinical judgement of the Investigator has a risk of suicide or has made a suicide attempt in the previous 12 months prior to the first dosing.
4. Positive urine drug or alcohol results at screening or at check-in.
5. Positive results at screening for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or antibody test for hepatitis C virus (HCV).
6. Unable to refrain from or anticipates the use of:

   * Any vaccines, drugs, including prescription and non-prescription medications, herbal remedies, or vitamin supplements within 14 days prior to the first dosing. Thyroid hormone replacement medication may be permitted if the participant has been on the same stable dose for the immediate 3 months prior to first dosing.
   * Any drugs known to be significant inducers of cytochrome P450 (CYP)3A, CYP2C19, uridine 5' diphospho-glucuronosyltransferase (UGT)1A9 or (UGT)2B4 enzymes and/or P-glycoprotein (P-gp), including St. John's Wort, within 28 days prior to the first dosing. Appropriate sources (example, Flockhart TableTM) will be consulted to confirm lack of Pharmacokinetics (PK)/pharmacodynamics interaction with study drug.
7. Consumes excessive amounts, defined as greater than 4 servings (1 serving is approximately equivalent to 120 mg of caffeine) of coffee, tea, cola, energy drinks or other caffeinated beverages per day.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10-11 (Estimated); Primary Completion 2022-12-06 (Estimated); Study Completion 2022-12-06 (Estimated)

PRIMARY OUTCOMES:
Placebo-corrected Change From Baseline in Corrected QT Interval (QTc) | Day -1 up to 24 hours post-dose
  The QTc interval will be measured by continuous electrocardiogram (ECG) recordings. The primary QT correction method will be Fridericia's correction. In case a substantial HR effect is observed on-treatment with soticlestat, drug-free QT/RR data will be collected over a range of Heart Rate (HR) seen off-treatment to allow the generation of individualized QT correction methods. QTc will be calculated from Day -1 of the first treatment period both during the periods of supine rest (QTcS) and from all evaluable QT/RR pairs in the 24-hour recording (QTcI). The method that removes the HR dependence of the QT interval most efficiently will be chosen as primary correction method. The analysis for QTc will be based on a linear mixed-effects model with ΔQTc as the dependent variable, period, sequence, time (that is, nominal post-dose time point), treatment, and time-by-treatment interaction as fixed effects, and baseline QTc as a covariate.

SECONDARY OUTCOMES:
Change From Baseline in HR | Day 1: Pre-dose up to 24 hours post-dose
  HR will be measured by continuous ECG recordings.
Change From Baseline in QTc With the Methods Not Selected as Primary | Day 1: Pre-dose up to 24 hours post-dose
  The QTc interval will be measured by continuous ECG recordings. Pre-dose will be the average of the derived ECG intervals from the 3 ECG time-points (-0.75, -0.5, and -0.25 hours) prior to treatment administration on Day 1 within each respective period.
Change From Baseline in Individualized HR-corrected QT interval (QTcS) | Day 1: Pre-dose up to 24 hours post-dose
  The QTcS interval will be measured by continuous ECG recordings and QT/RR interval of ECG (RR) data obtained at supine resting time points. The analysis for QTcS will be based on a linear mixed-effects model.
Change From Baseline in Optimized QT Interval (QTcI) | Day 1: Pre-dose up to 24 hours post-dose
  The QTcI interval will be measured by continuous ECG recordings and QT/RR data obtained at supine resting time points. The analysis for QTcI will be based on a linear regression model.
Change From Baseline in PR Interval of the ECG (PR) | Day 1: Pre-dose up to 24 hours post-dose
  PR will be measured by continuous ECG recordings.
Change From Baseline in QRS Interval of the ECG (QRS) | Day 1: Pre-dose up to 24 hours post-dose
  QRS will be measured by continuous ECG recordings.
Placebo-corrected Change From Baseline in HR | Day 1: Pre-dose up to 24 hours post-dose
  Placebo-corrected HR will be measured by continuous ECG recordings.
Placebo-corrected Change From Baseline in QTc With the Methods Not Selected as Primary | Day 1: Pre-dose up to 24 hours post-dose
  Placebo-corrected QTc interval will be measured by continuous ECG recordings. Pre-dose will be the average of the derived ECG intervals from the 3 ECG time-points (-0.75, -0.5, and -0.25 hours) prior to treatment administration on Day 1 within each respective period.
Placebo-corrected Change From Baseline in PR Interval of ECG | Day 1: Pre-dose up to 24 hours post-dose
  Placebo-corrected PR interval will be measured by continuous ECG recordings.
Placebo-corrected Change From Baseline in QRS Interval of ECG | Day 1: Pre-dose up to 24 hours post-dose
  Placebo-corrected QRS interval will be measured by continuous ECG recordings.
Number of Participants with Categorical Outlier Values for HR | Day 1: Pre-dose up to 24 hours post-dose
  Number of participants with categorical outlier values for HR will be determined. A participant will be determined as an outlier if the following criteria were met for the ECG intervals at any time point: Decrease of HR from baseline greater than (>) 25 percent (%) resulting in HR less than (<) 50 beats per minute (bpm) and increase in HR from baseline resulting in HR >100 bpm.
Number of Participants with Categorical Outliers Values for PR | Day 1: Pre-dose up to 24 hours post-dose
  Number of participants with categorical outlier values for PR will be determined. A participant will be determined as an outlier if the following criteria were met for the ECG interval at any time point: Increase of PR from Baseline >25% resulting in PR >200 millisecond (ms).
Number of Participants with Categorical Outliers Values for QRS | Day 1: Pre-dose up to 24 hours post-dose
  Number of participants with categorical outliers values for QRS will be determined. A participant will be determined as an outlier if the following criteria were met for the ECG interval at any time point: Increase of QRS from Baseline >25% resulting in QRS >120 ms.
Number of Participants with Categorical Outliers Values for QTc | Day 1: Pre-dose up to 24 hours post-dose
  Number of participants with categorical outliers values for QTc will be determined. A participant will be determined as an outlier if the following criteria were met for the ECG interval at any time point: Increase in treatment-emergent value >450 and less than or equal to (<=) 480 ms; >480 and <=500; change from Baseline of >30 and <=60 ms or >60 ms.
Percentage of Participants with Change From Baseline in ECG Morphology | Day 1: Pre-dose up to 24 hours post-dose
  ECG morphological analyses will be performed using the ECG waveform interpretation as defined by the central ECG laboratory's cardiologist.
Number of Participants Reporting one or More Treatment-emergent Adverse Events (TEAEs) | Baseline (Day 1) up to 14 days after the last dose of study drug in Period 4 (Day 39)
  An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant who has signed informed consent to participate in a study; it does not necessarily have to have a causal relationship with the treatment. A TEAE is defined as an adverse event with an onset that occurs after receiving study drug.
Cmax: Maximum Observed Plasma Concentration for Soticlestat | Day 1: Pre-dose and at multiple timepoints (up to 24 hours) post-dose
AUC∞: Area Under the Plasma Concentration-time Curve from Time 0 to Infinity for Soticlestat | Day 1: Pre-dose and at multiple timepoints (up to 24 hours) post-dose
AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Soticlestat | Day 1: Pre-dose and at multiple timepoints (up to 24 hours) post-dose
Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Soticlestat | Day 1: Pre-dose and at multiple timepoints (up to 24 hours) post-dose
T1/2z: Terminal Phase Elimination Half-life for Soticlestat | Day 1: Pre-dose and at multiple timepoints (up to 24 hours) post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/2089cfe856aa4315?idFilter=%5B%22TAK-935-1001%22%5D